CLINICAL TRIAL: NCT04311762
Title: Phase 1 Trial of Endobronchial Ultrasound-Guided Transbronchial Needle Injection of Cisplatin for Stage IV Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, C. Matthew Kinsey MD, MPH, Director, Interventional Pulmonary, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00000613
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer Metastatic
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Initial Treatment- Low Perfusion Region (Experimental): Phase 1B uses a within group comparison. All participants will undergo 1 delivery of intratumoral cisplatin into either a low or high perfusion region, then the subsequent week undergo delivery into the other region, for a total of 3 treatments.
  Interventions: Drug: cisplatin

INTERVENTIONS:
Drug: cisplatin — Intratumoral delivery of cisplatin via bronchoscopy (endobronchial ultrasound)
  Other Names: Platinol

SUMMARY:
The goal of the study is to identify the maximum tolerated dose of endobronchial ultrasound-guided transbronchial injection (EBUS-TBNI) of cisplatin for Stage IV lung cancer.

DETAILED DESCRIPTION:
Multiple studies have demonstrated feasibility and safety of delivering cisplatin directly into lung tumors using endobronchial ultrasound guided-transbronchial needle injection (EBUS-TBNI). This technique relies on the use of a bronchoscope with an integrated ultrasound transducer allowing real-time visualization of, and delivery of cisplatin into, tumors lying in proximity to the central airways. Prior work has utilized this technique to treat loco regional recurrence in a previously radiated field. The goal of the current study is to identify the initial dose for intratumoral cisplatin. Phase 1A is a dose ranging study. Phase 1B is designed to evaluate the safety of delivery of the drug into different tumor regions .

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or above

Eastern Cooperative Oncology Group (ECOG) performance score 0-2

Have known or suspected metastatic NSCLC at time of enrollment (including patients who progress on initial therapy or are found to have metastatic disease during therapy and are not excluded based on 8.2 below).

Ability and willingness to provide informed consent

A CT scan of the chest (with or without contrast) within the prior 3 months.

The presence of an EBUS accessible target site. These may be primary lung cancers or metastatic sites (including when a lymph node station has been replaced by metastatic tumor), that are accessible by EBUS

Patients must have adequate organ and marrow function as defined below:

* Leukocytes ≥3,000/mcL
* Platelets ≥100,000/mcL
* Total bilirubin ≤ institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) ≤ institutional ULN
* Glomerular filtration rate (GFR) ≥60 mL/min/1.73 m2 via CKD EPI)

Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

Exclusion Criteria:

Use of an investigational agent in prior 30 days

Pregnancy/lactation

Treatment with cytotoxic chemotherapy within the past 30 days

Prior (within the last 12 months) or ongoing radiation treatment to the study NSCLC

Allergy to cisplatin or its derivatives

Patient not appropriate for the research study based on physician discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: C. Matthew Kinsey, MD, MPH, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No